CLINICAL TRIAL: NCT03194386
Title: Feasibility and Interest of Early Eye-Movement Desensitization and Reprocessing Provided in the Emergency Department for Patients With High Risk of Post Traumatic Syndrome
Brief Title: Eye-Movement Desensitization and Reprocessing in the ED and Post-Traumatic Syndrome
Acronym: EMDR-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017/01
Record Dates: First submitted 2017-03-24; First posted 2017-06-21 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2017-06

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Post-Traumatic Syndrome; Eye-Movement Desensitization and Reprocessing
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigator / Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): usual care
- Reassurance (Active Comparator): 15 minutes psychologist visit
  Interventions: Other: Reassurance
- R-TEP EMDR (Experimental): Recent Traumatic Episode Protocol Eye-Movement Desensitization and Reprocessing (R-TEP EMDR) At the end of cares, before ED discharge, a trained psychologist will conduct a single R-TEP EMDR session. Each session may last about 60 minutes
  Interventions: Other: Eye-Movement Desensitization and Reprocessing (EMDR)

INTERVENTIONS:
Other: Reassurance — At the end of cares, before ED discharge, a trained psychologist will conduct a session in order to reassure patients about their future after ED visit.
  Arms: Reassurance
Other: Eye-Movement Desensitization and Reprocessing (EMDR) — At the end of cares, before ED discharge, a trained psychologist will conduct a single EMDR session. Each session may last about 60 minutes
  Arms: R-TEP EMDR

SUMMARY:
Millions people, all over the world, are admitted in the Emergency Department after a trauma or simply to receive medical cares. In France, it represents 10 million patients. Probably because of stress associated with the event, 20% will suffer a combination of non-specifics symptoms which persist for many months and with daily life quality impairment. The investigators hypothesize that an early intervention, such as Eye-Movement, Desensitization and Reprocessing (EMDR) could be performed in the ED and could prevent the occurrence of these symptoms

DETAILED DESCRIPTION:
Emergency department are a privileged service for patients suffering from trauma and stressful medical conditions. In France every year 10 million people come or are taken to the emergency room (ER). Many studies have shown that 10-20% of these trauma patients develop a non-specific set of symptoms that can persist for several months after ED assessment. These includes, for example, headache, memory and/or concentration impairment, stress intolerance, irritability... These symptoms lead to an alteration in the quality of social, family and professional life, and therefore affect one to two millions people in France alone.

The association between these symptoms and mild traumatic brain injury (MTBI) has already been demonstrated. It was defined as post-concussion syndrome (PCS) according to the DSM-IV-TR. However, several recent studies have shown that these symptoms are not specific to MTBI but may appear for any type of trauma and event for stressful medical conditions. PCS seems to appear for events occurring in a stressful environment or in people with psychological weaknesses. These symptoms will therefore be referred here to PCS-like syndrome (PCSLS). Moreover, PCS-LS symptoms appear to be very similar to those of the numbing and hyperarousal dimension of the Post Traumatic Stress Disorder (PTSD).

A recent study, carried out by our team in the ED of Bordeaux University Hospital, showed that PCS-LS was associated with a high level of stress at ED discharge, whatever that stress level at entry.

The Eye-Movement Desensitization and Reprocessing (EMDR) is a recognized psychotherapeutic approach in the treatment of PTSD and several single-session versions of the protocol have been proposed (R-TEP EMDR).The investigators hypothesize that the introduction of an early R-TEP EMDR intervention in emergencies can reduce the level of stress and thus the occurrence of the PCSLS and PTSD symptoms among a subset of patients screened for their high risk of PCS-LS.

The study is a single-site open-label three-group randomized controlled trial designed to assess the feasibility of an early R-TEP EMDR intervention performed in the ED and to compare PCS-LS and PTSD symptoms at 3 months between the three randomization groups: (i) TEP-EMDR; (ii) 15' reassurance session; (iii) care as usual.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in department for a medical or traumatic event, and at risk of developing a PTS.
* Score resulting from the screening tool> 3 :

Female gender: +1 Taking at least one anxiolytic treatment: + 1 Perceived health status prior to admission: Excellent, very good: 0 ; Good: +1 Poor: +2 ; Bad: +3

* Affiliated to Social Security

Exclusion Criteria:

* Refusal to participate in the study
* Admission and / or exit questionnaire not completed
* Inability to answer questionnaire: any cognitive impairement, language barrier, consciousness disorder...
* Impossibility of recontacting the patient at a distance from the trauma (no telephone contact ...)
* Patient already included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
EMDR protocol completion | 12 hours after ED admission
  Eye-Movement Desensitization and Reprocessing, performed in a population with high risk of PTS at the Emergency Department thanks to questionnaires

SECONDARY OUTCOMES:
Recovery rate | 3 months
  3 months after ED admission
Post-concussion Syndrome | 3 months after ED admission
  Post-Concussion Syndrome (PCS) was assessed using the various definitions of PCS (ICD-10, DSM IV and Rivermaid) were selected: headache, feelings of dizziness, nausea or vomiting, noise sensitivity, sleeping disorders, fatigue, irritability, feeling depressed, anxiety, intolerance to stress, feeling frustrated or impatient, forgetfulness or poor memory, poor concentration, taking longer to think, blurred vision, double vision, light sensitivity, restlessness, personality change. In line with PCS definition in the context of mild head injury, we defined patients with PCS as those who reported at least 3 of these symptoms.
Post-Traumatic Stress Disorder | 3 months after ED admission
  Post-Traumatic Stress Disorder was defined using the PTSD Check-List Scale. The presence of the 17 symptoms of the DSM-IV-R definition for PTSD were also assessed for the 3-month phone The diagnosis of PTSD requires that one or more symptoms from each of those categories be present for at least a month and that those symptoms interfere seriously with leading a normal life.
Chronic Pain at 3 months | 3 months after ED admission
  Self reported by phone

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Lagarde, PhD, Study Director — University Hospital Bordeaux, France
Locations (1):
- Emergency department, Bordeaux University Hospital, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Gil-Jardine C, Evrard G, Al Joboory S, Tortes Saint Jammes J, Masson F, Ribereau-Gayon R, Galinski M, Salmi LR, Revel P, Regis CA, Valdenaire G, Lagarde E. Emergency room intervention to prevent post concussion-like symptoms and post-traumatic stress disorder. A pilot randomized controlled study of a brief eye movement desensitization and reprocessing intervention versus reassurance or usual care. J Psychiatr Res. 2018 Aug;103:229-236. doi: 10.1016/j.jpsychires.2018.05.024. Epub 2018 May 26. PMID 29894921